CLINICAL TRIAL: NCT02434380
Title: Effect of Vitamin D Replacement on Maternal and Neonatal Outcomes: a Randomized Controlled Trial in Pregnant Women With Hypovitaminosis D
Brief Title: Effect of Vitamin D Replacement on Maternal and Neonatal Outcomes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: American University of Beirut Medical Center (Other)
Collaborators: University of Southampton (Other); Bahman Hospital Beirut Lebanon (Unknown)
Responsible Party: Principal Investigator, Dr. Ghada El-Hajj Fuleihan, Professor of Medicine, American University of Beirut Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AUBMC-GE-HF-2; AUBMC-IM-GE-HF-22 (Other Grant/Funding Number: American University of Beirut)
Record Dates: First submitted 2015-04-27; First posted 2015-05-05 (Estimated); Last update posted 2023-03-20 (Actual); Status verified 2023-03

CONDITIONS: Hypovitaminosis D; Pregnancy Complications; Infant, Newborn, Diseases
Keywords: Vitamin D; Bone mineral content; Knee-heel length; Middle East
MeSH Terms: conditions — Vitamin D Deficiency; Pregnancy Complications; Infant, Newborn, Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Low dose vitamin D (Active Comparator): Vitamin D3 Euro D 10,000 IU (1 tablet) plus Euro D Placebo (1 tablet) weekly, alternating with Euro D Placebo (2 tablets) weekly, starting at the second trimester and continued until delivery.
  Interventions: Dietary Supplement: Euro D
- High dose vitamin D (Active Comparator): Vitamin D3 Euro D 10,000 IU (2 tablets, equivalent to 20,000 IU) weekly, starting at the second trimester and continued until delivery.
  Interventions: Dietary Supplement: Euro D

INTERVENTIONS:
Dietary Supplement: Euro D — Vitamin D3 Euro D 10,000 IU (1 tablet) plus Euro D Placebo (1 tablet) weekly, alternating with Euro D Placebo (2 tablets) weekly, starting at the second trimester and continued until delivery.
  Other Names: Europharm
  Arms: Low dose vitamin D
Dietary Supplement: Euro D — Vitamin D3 Euro D 10,000 IU (2 tablets, equivalent to 20,000 IU) weekly, starting at the second trimester and continued until delivery.
  Other Names: Europharm
  Arms: High dose vitamin D

SUMMARY:
The optimal vitamin D replacement dose during pregnancy remains undefined. Therefore, the aim of this study is to test the hypothesis that a daily equivalent dose of vitamin D of 3,000 IU/day is needed for Middle Eastern women, to optimize maternal vitamin D level and neonatal musculoskeletal parameters, specifically knee-heel length at birth and bone mineral content at one month of age.

DETAILED DESCRIPTION:
Hypovitaminosis D is prevalent worldwide across the lifecycle, including pregnant women, and particularly in the Middle East. It has been associated with adverse maternal and neonatal outcomes. While the Institute of Medicine (IOM) recommends 600 IU of vitamin D per day to reach a 25-Hydroxyvitamin D (25(OH)D) level ≥ 20 ng/ml, the Endocrine Society (ES) recommends 1,500-2,000 IU/day to reach a level ≥ 30 ng/ml, and the WHO guidelines do not recommend any supplementation as part of routine prenatal care. They do however underscore the fact that subjects with the lowest levels may be the ones to benefit most from vitamin D replacement. The benefits of such an approach and the doses needed to reach desirable levels have not been tested. This randomized trial proposes to do so, testing the effect of two vitamin D doses, a low dose of 600 IU daily and a high dose of 3,000 IU daily.

330 pregnant women, with 25(OH)D level 10-30 ng/ml during the early second trimester will be recruited form the American University of Beirut-Medical Center (AUB-MC), and Bahman Hospital. They will be randomized, in a double blinded fashion, to receive daily equivalent doses of cholecalciferol, 600 IU or 3,000 IU until delivery. Maternal clinical information and a food frequency questionnaire will be obtained at each visit until delivery. Maternal 25(OH)D and chemistries, including Calcium, creatinine, lipid profile, glucose and Insulin will be assessed at study entry, during third trimester and at delivery. Fetal measurements will be collected at study entry and during the second trimester. Neonatal anthropometric variables and venous umbilical cord 25(OH)D level will be measured at birth and infants will also undergo dual-energy x-ray absorptiometry (DEXA) scan assessment, for bone and fat mass, at one to 6 weeks. Maternal and neonatal genetic studies for vitamin D genes polymorphism, and other modules of placnetal calcium transport will be also performed.

Throughout the study, adverse events will be collected systematically and an independent Data and Safety Monitoring Board will be asked to review serious adverse events.

The percent of women achieving 25(OH)D ≥ 20ng/ml in the low dose will be compared to that in the high dose using Chi-Square. Independent t-test will be used to compare mean neonatal bone mineral content at one month of age between the 2 arms. For other outcomes, t-test will be used for continuous outcomes and Chi-square will be used for binary outcomes to compare means and proportions, respectively. The primary analysis is an intention-to-treat analysis (ITT) of unadjusted results. For the primary outcomes, p- values will be considered statistically significant if ≤ 0.025.

The investigators study would be the only randomized controlled trial in the Middle East, to investigate the recommended daily allowance for vitamin D, and the desirable dose to optimize neonatal musculoskeletal health, in women with low 25(OH)D levels, levels that are reflective of those in most countries from the Middle East.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women gestational age (GA)< 14 weeks at screening visit. Middle Eastern woman (Middle East countries defined by WHO: Bahrain, Egypt, Iran, Iraq, Palestine, Jordan, Kuwait, Lebanon, Oman, Qatar, Saudi Arabia, Syria, , United Arab Emirates, Yemen)
* 25(OH)D level between 10ng/ml and 30ng/ml
* Age > 18 years
* Vitamin D supplementation ≤ 200 IU daily (If daily vitamin D supplementation > 200 IU daily, at enrollment, the pregnant women will be advised to adjust prenatal multivitamin doses in such a way that total vitamin D supplementation per week doesn't exceed 1400 IU per week, in consultation with primary Obstetric and Gynecology (OB-GYN) physician.)

Exclusion Criteria:

* 25(OH)D level < 10 ng/ml or > 30 ng/ml.
* Known metabolic bone disease
* Current medications likely to interfere with vitamin D metabolism (enzyme inducing anticonvulsants, anti -TB)
* Vitamin D supplementation > 600 IU daily
* Pregnant women with twins

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 330 (Estimated)
Dates: Start 2015-07; Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
The proportions of women who will reach the IOM defined desirable 25(OH)D level ≥20ng/ml. | At delivery
Infant bone mineral content (BMC) | one to six weeks
  We will assess Infant bone mineral content (BMC) by whole body dual-energy x-ray absorptiometry (DEXA) scan

SECONDARY OUTCOMES:
Maternal 25(OH)D level | At delivery
  We will assess mean maternal 25(OH)D level
Neonatal 25(OH)D level, at delivery | At birth
  We will assess mean neonatal 25(OH)D level
Mean infant fat mass | At one month of age
  We will assess Infant fat mass by whole body dual-energy x-ray absorptiometry (DEXA) scan
Neonatal Knee to heel length at birth | At birth
  We will assess neonatal Knee to heel length at birth using simple vernier calipers
Maternal Parathyroid Hormone (PTH) Level | At delivery
  We will assess mean maternal PTH level
Neonatal Parathyroid Hormone (PTH) Level | At birth
  We will assess mean neonatal PTH level
Mean change in maternal urine calcium | Change between baseline and 3 months following intervention
  We will assess the change in urine calcium level after 3 months of vitamin D supplementation.

OTHER OUTCOMES:
Composite outcome (incidence of C-section and gestational diabetes mellitus (GDM)) | At delivery
  We will assess the incidence of a composite outcome (C-section and gestational diabetes mellitus (GDM)) in a subgroup of women who has no previous C-section.
Maternal weight | At delivery
Maternal Blood Pressure (BP) | At delivery
Number of ill days | At 28-32 weeks Gestational Age (GA) and at delivery
Intrauterine fetal skeletal measures | At 11-13 weeks and at 20 weeks
  We will collect intrauterine fetal skeletal measures including crown-rump, femur length, abdominal circumference, head circumference, biparietal diameter
APGAR score | At delivery
  Proportion of neonates with low APGAR (<7) score at 1 and 5 minutes, at delivery
Neonatal weight | At birth
Neonatal length | At birth
Placental weight | At delivery
Placental 1α hydroxylase activity | At delivery
Sub-group analysis: The proportions of women who will reach the IOM defined desirable 25(OH)D level ≥20ng/ml. | At delivery
  Subgroup analysis based on baseline 25(OH)D, less than 20 ng/ml versus less than 30 ng/ml and season of birth will be performed
Sub-group analysis:Infant bone mineral content (BMC) | One month of age
  Subgroup analysis based on baseline 25(OH)D, less than 20 ng/ml versus less than 30 ng/ml and season of birth will be performed.

CONTACTS AND LOCATIONS:
Overall Officials: Ghada El Hajj Fuleihan, Professor of Medicine, Principal Investigator — American University of Beirut Medical Center
Locations (1):
- American University of Beirut, Hamra, Lebanon

REFERENCES:
- [Background] Kovacs CS, Fuleihan Gel-H. Calcium and bone disorders during pregnancy and lactation. Endocrinol Metab Clin North Am. 2006 Mar;35(1):21-51, v. doi: 10.1016/j.ecl.2005.09.004. No abstract available. PMID 16310641
- [Background] Bassil D, Rahme M, Hoteit M, Fuleihan Gel-H. Hypovitaminosis D in the Middle East and North Africa: Prevalence, risk factors and impact on outcomes. Dermatoendocrinol. 2013 Apr 1;5(2):274-98. doi: 10.4161/derm.25111. PMID 24194968
- [Background] Arabi A, El Rassi R, El-Hajj Fuleihan G. Hypovitaminosis D in developing countries-prevalence, risk factors and outcomes. Nat Rev Endocrinol. 2010 Oct;6(10):550-61. doi: 10.1038/nrendo.2010.146. PMID 20852586
- [Background] Mithal A, Wahl DA, Bonjour JP, Burckhardt P, Dawson-Hughes B, Eisman JA, El-Hajj Fuleihan G, Josse RG, Lips P, Morales-Torres J; IOF Committee of Scientific Advisors (CSA) Nutrition Working Group. Global vitamin D status and determinants of hypovitaminosis D. Osteoporos Int. 2009 Nov;20(11):1807-20. doi: 10.1007/s00198-009-0954-6. Epub 2009 Jun 19. PMID 19543765
- [Background] Hoteit M, Al-Shaar L, Yazbeck C, Bou Sleiman M, Ghalayini T, Fuleihan Gel-H. Hypovitaminosis D in a sunny country: time trends, predictors, and implications for practice guidelines. Metabolism. 2014 Jul;63(7):968-78. doi: 10.1016/j.metabol.2014.04.009. Epub 2014 Apr 23. PMID 24874590
- [Background] El-Hajj Fuleihan G, Nabulsi M, Tamim H, Maalouf J, Salamoun M, Khalife H, Choucair M, Arabi A, Vieth R. Effect of vitamin D replacement on musculoskeletal parameters in school children: a randomized controlled trial. J Clin Endocrinol Metab. 2006 Feb;91(2):405-12. doi: 10.1210/jc.2005-1436. Epub 2005 Nov 8. PMID 16278262
- [Background] Morley R, Carlin JB, Pasco JA, Wark JD. Maternal 25-hydroxyvitamin D and parathyroid hormone concentrations and offspring birth size. J Clin Endocrinol Metab. 2006 Mar;91(3):906-12. doi: 10.1210/jc.2005-1479. Epub 2005 Dec 13. PMID 16352684
- [Background] Al-Shaar L, Mneimneh R, Nabulsi, Maalouf J, Fuleihan Gel-H. Vitamin D3 dose requirement to raise 25-hydroxyvitamin D to desirable levels in adolescents: results from a randomized controlled trial. J Bone Miner Res. 2014 Apr;29(4):944-51. doi: 10.1002/jbmr.2111. PMID 24123134
- [Background] Parkes I, Schenker JG, Shufaro Y. Parathyroid and calcium metabolism disorders during pregnancy. Gynecol Endocrinol. 2013 Jun;29(6):515-9. doi: 10.3109/09513590.2012.754880. Epub 2013 Jan 25. PMID 23350730
- [Background] Nassar N, Halligan GH, Roberts CL, Morris JM, Ashton AW. Systematic review of first-trimester vitamin D normative levels and outcomes of pregnancy. Am J Obstet Gynecol. 2011 Sep;205(3):208.e1-7. doi: 10.1016/j.ajog.2011.03.058. Epub 2011 Apr 7. PMID 21640968
- [Background] Hollis BW, Wagner CL. Vitamin D and pregnancy: skeletal effects, nonskeletal effects, and birth outcomes. Calcif Tissue Int. 2013 Feb;92(2):128-39. doi: 10.1007/s00223-012-9607-4. Epub 2012 May 24. PMID 22623177
- [Background] Thorne-Lyman A, Fawzi WW. Vitamin D during pregnancy and maternal, neonatal and infant health outcomes: a systematic review and meta-analysis. Paediatr Perinat Epidemiol. 2012 Jul;26 Suppl 1(0 1):75-90. doi: 10.1111/j.1365-3016.2012.01283.x. PMID 22742603
- [Background] Harvey NC, Moon RJ, Sayer AA, Ntani G, Davies JH, Javaid MK, Robinson SM, Godfrey KM, Inskip HM, Cooper C; Southampton Women's Survey Study Group. Maternal antenatal vitamin D status and offspring muscle development: findings from the Southampton Women's Survey. J Clin Endocrinol Metab. 2014 Jan;99(1):330-7. doi: 10.1210/jc.2013-3241. Epub 2013 Dec 20. PMID 24178796
- [Background] Javaid MK, Crozier SR, Harvey NC, Gale CR, Dennison EM, Boucher BJ, Arden NK, Godfrey KM, Cooper C; Princess Anne Hospital Study Group. Maternal vitamin D status during pregnancy and childhood bone mass at age 9 years: a longitudinal study. Lancet. 2006 Jan 7;367(9504):36-43. doi: 10.1016/S0140-6736(06)67922-1. PMID 16399151
- [Background] Ross AC, Manson JE, Abrams SA, Aloia JF, Brannon PM, Clinton SK, Durazo-Arvizu RA, Gallagher JC, Gallo RL, Jones G, Kovacs CS, Mayne ST, Rosen CJ, Shapses SA. The 2011 report on dietary reference intakes for calcium and vitamin D from the Institute of Medicine: what clinicians need to know. J Clin Endocrinol Metab. 2011 Jan;96(1):53-8. doi: 10.1210/jc.2010-2704. Epub 2010 Nov 29. PMID 21118827
- [Background] Holick MF, Binkley NC, Bischoff-Ferrari HA, Gordon CM, Hanley DA, Heaney RP, Murad MH, Weaver CM; Endocrine Society. Evaluation, treatment, and prevention of vitamin D deficiency: an Endocrine Society clinical practice guideline. J Clin Endocrinol Metab. 2011 Jul;96(7):1911-30. doi: 10.1210/jc.2011-0385. Epub 2011 Jun 6. PMID 21646368
- [Background] Harvey N, Dennison E, Cooper C. Osteoporosis: a lifecourse approach. J Bone Miner Res. 2014 Sep;29(9):1917-25. doi: 10.1002/jbmr.2286. PMID 24861883
- [Background] De-Regil LM, Palacios C, Ansary A, Kulier R, Pena-Rosas JP. Vitamin D supplementation for women during pregnancy. Cochrane Database Syst Rev. 2012 Feb 15;2(2):CD008873. doi: 10.1002/14651858.CD008873.pub2. PMID 22336854
- [Background] Hollis BW, Johnson D, Hulsey TC, Ebeling M, Wagner CL. Vitamin D supplementation during pregnancy: double-blind, randomized clinical trial of safety and effectiveness. J Bone Miner Res. 2011 Oct;26(10):2341-57. doi: 10.1002/jbmr.463. Erratum In: J Bone Miner Res. 2011 Dec; 26(12):3001. PMID 21706518
- [Background] Dawodu A, Saadi HF, Bekdache G, Javed Y, Altaye M, Hollis BW. Randomized controlled trial (RCT) of vitamin D supplementation in pregnancy in a population with endemic vitamin D deficiency. J Clin Endocrinol Metab. 2013 Jun;98(6):2337-46. doi: 10.1210/jc.2013-1154. Epub 2013 Apr 4. PMID 23559082
- [Derived] Assaad M, Fuleihan GE, Nassar A, MScs SA, MScs MR, Cooper C, Harvey NC, Tfaily N, Diab T, Al-Tayeh R, Chakhtoura M. Enhancing the Implementation of a high-quality randomized trial in pregnancy. Res Sq [Preprint]. 2026 Jan 12:rs.3.rs-8287988. doi: 10.21203/rs.3.rs-8287988/v1. PMID 41646349
- [Derived] Chakhtoura M, Nassar A, Arabi A, Cooper C, Harvey N, Mahfoud Z, Nabulsi M, El-Hajj Fuleihan G. Effect of vitamin D replacement on maternal and neonatal outcomes: a randomised controlled trial in pregnant women with hypovitaminosis D. A protocol. BMJ Open. 2016 Mar 8;6(3):e010818. doi: 10.1136/bmjopen-2015-010818. PMID 26956166
- See also: Calcium Metabolism and Osteoporosis Program, American University of Beirut — http://website.aub.edu.lb/fm/cmop/Pages/Publications.aspx